CLINICAL TRIAL: NCT06168994
Title: Role of Eplerenone in Reducing Recurrence of Atrial Fibrillation in Patient With Structural Heart Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walid Shehata Ahmed abdellah, Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Eplerenone in AF
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiodarone as comparison (Active Comparator): 50 patients >>Amiodarone +other treatmen
  Interventions: Drug: Eplerenone
- Eplerenone plus amiodarone (Experimental): 50 patients >>Amiodarone +other treatmen
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — Amiodarone vs eplerenone in AF

SUMMARY:
The aim of this study is to study synergistic effect of eplerenone as Selective aldosterone receptor antagonist with amiodarone compared with amiodarone only in reducing recurrence of atrial fibrillation in patient with structural heart disease

DETAILED DESCRIPTION:
Atrial fibrillation is the most common sustained arrhythmia, with a rising prevalence that substantially increases the risk of stroke and heart failure (1,2), The rate of recurrences without antiarrhythmic treatment is 71%-84%, and it can be reduced to 44%-67% with antiarrhythmic drug therapy(3) Mineralocorticoid receptor blockers (MRBs) are beneficial in systolic HF[ 4,5,6]. Specifically, the MRB eplerenone (EPL) has been shown to reduce new onset AF and recurrent AF in HF patients (7). Both angiotensin II and aldosterone elevations may lead to atrial fibrosis and contribute to human AF (8). Experimental results suggest that aldosterone may cause a substrate for atrial fibrosis and AF (9). Aldosterone increases the expression of 11β-hydroxysteroid dehydrogenase type 2 (11b-HSD2) leading to up-regulation of profibrotic mediators and collagen synthesis, which is prevented by MRBs (10).

The European Society of Cardiology (ESC) guidelines identify AF as secondary to Structural heart diseases (SHDs)when a left ventricle (LV) systolic or diastolic dysfunction is demonstrated or LV hypertrophy, valvular disease, and/or other SHDs are documented [11].currently, SHD includes: (a) heart failure with reduced ejection fraction (HFrEF, previously severe or moderate LV systolic dysfunction); (b) heart failure with preserved ejection fraction (HFpEF, previously LV diastolic dysfunction); (c) valvular heart disease (VHD) and (d) specific cardiomyopathies, such as hypertrophic cardiomyopathy (HCM) [12].

Electrical remodelling is the first mechanism that occurs at the onset of AF and promotes AF through a re-entry-prone substrate. Changes in atrial frequency are determined by changes in the physiology of ion channel activation[13] Amiodarone is an antiarrhythmic medication used to treat and prevent a number of types of cardiac dysrhythmias,it blocks the channels that are upregulated by remodelling such as inward-rectifying K1 current (IK1) or by stimulation of the sympathetic nervous system.[14]

ELIGIBILITY:
Inclusion Criteria:

- paroxysmal AF who reverted to sinus rhythm either medically or electrically without appropriate secondary cause of primary AF

•AF attack should be documented with ECG

Exclusion Criteria:

* 1-patients are currently on eplerenone or spironolactone 2-hyperkalemia 3-impaired renal function(if CrCl <50ml/min or serum creatinine>2 mg/dl) 4-patient on beta blocker and calcium channel blocker (non- dihydropyridine) 5-prosthetic valve 6-severe mitral stenosis 7-thyroid dysfunction 8-WPW 9-severe liver disease 10-persistent or permanent AF 11-pregnancy or breast feeding 12-LV EF<50% 13-known hypersensitivity or drug reaction to amiodarone 14-acute coronary syndrome 15-refusal of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2026-09-29 (Estimated); Study Completion 2027-05-20 (Estimated)

PRIMARY OUTCOMES:
Role of eplerenone in reducing recurrence of atrial fibrillation in patient with structural heart disease | Baseline
  decrease recurrence of paroxysmal AF in patient of structural heart disease